CLINICAL TRIAL: NCT03706703
Title: The Safety and Efficacy of Rh-Endostatin (Endostar®) Continuous Intravenous Infusion in Combination With Docetaxel/Carboplatin or Pemetrexed/Carboplatin (DC/PC) Regimens for Untreated Stage IIIB/IV Non-small-cell Lung Cancer (NSCLC)
Brief Title: Rh-Endostatin (Endostar®) Continuous Intravenous Infusion
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Affiliated Cancer Hospital & Institute of Guangzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ENDOSTAR
Record Dates: First submitted 2018-10-09; First posted 2018-10-16 (Actual); Last update posted 2018-10-17 (Actual); Status verified 2018-10

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — endostar protein; Docetaxel; Carboplatin; Pemetrexed

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Endostar continuous intravenous infusion (Experimental): Endostar continuous intravenous infusion in combination with docetaxel/carboplatin or pemetrexed/carboplatin
  Interventions: Drug: Endostar; Drug: Docetaxel; Drug: Carboplatin; Drug: Pemetrexed

INTERVENTIONS:
Drug: Endostar — continuous intravenous infusion Endostar,7.5mg/m2, continuous intravenous infusion for 14 days each cycle, 21 days as one cycle, 4 cycles in total.
Drug: Docetaxel — docetaxel is 75 mg/m2 intravenously over 1 hour on Day 1 of each 21-day cycle
Drug: Carboplatin — carboplatin is administered on Day 1 of each 21-day，followed by docetaxol or pemetrexed
Drug: Pemetrexed — pemetrexed is 500 mg/m2 intravenously on Days 1 of each 21-day cycle

SUMMARY:
Endostar is a anti-angiogenesis product and has been launched in China . The efficacy and safety have been defined. However, the compliance is unsatisfactory since routine i.v of Endostar is needed for 3 to 4 hours daily during one cycle of 14 days. The continuous intravenous infusion by using venous pump can improve the compliance.

ELIGIBILITY:
Inclusion criteria:

Primary non-small cell lung cancer confirmed by cytology and histology, excluding sputum examination;

Phase IIIB/IV based on TNM criteria (8th);

At least one measurable tumor based on RECIST 1.1;

Without the known active mutation of EGFR/ALK/ROS1/RET;

Male or female, age≥18 or ≤70 years old;

ECOG PS: 0 or 1;

Estimated time of survival: ≥ 3 months;

Suitable hematologic function: ANC≥2×109/L, PLC≥100×109/L and Hb≥9 g/dL;

Suitable liver function: Total bilirubin≤ normal ULN, AST and ALT≤2.5×normal ULN, ALP≤ 5×normal ULN;

Suitable renal function: Cr≤normal ULN,or Ccr≥60 ml/min;

EKG normal;

Without healing wound;

No history of anti-cancer therapy, or adjuvant/neo-adjuvant chemotherapy for non-metastatic tumor finished for more than 6 months before enrollment;

For the female subject with productive ability, urine pregnancy test must be done and is negative within 7 days before enrollment;

No history of serious allergic to biologic agents, especially E.Coli products;

The authorized ICF must be signed.

Exclusion Criteria:

Woman in pregnancy and breast-feeding, or having productive ability without contraception;

Having the serious acute infection uncontrolled or purulent/chronic infection with unhealed wound;

Having the serious heart disease, including congestive heart failure, uncontrolled high-risk arrhythmia, unstable angina, myocardial infarction, valvular disease, and refractory hypertension;

Having uncontrolled nervous or mental disease with low compliance and reluctance to description of response; uncontrolled primary brain tumor or other metastatic brain cancer with obvious intracranial hypertension or mental symptoms;

Having the tendency of bleeding, such as FIB≤2G/L;

Being receiving adjuvant chemotherapy;

On other conditions investigator considers, the subject is not fitful to participate the trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-04-01 (Estimated); Study Completion 2020-09-01 (Estimated)

PRIMARY OUTCOMES:
ORR | 8 weeks
  objective response rate based on Recist 1.1 edition

SECONDARY OUTCOMES:
PFS | 8 weeks
  progress free survival

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Cancer Hospital & Institute of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided